CLINICAL TRIAL: NCT06799052
Title: Same-Day Cervical Preparation Prior to Second Trimester Dilation & Evacuation: A Noninferiority Randomized Control Trial Comparing Single-Balloon Catheter and Osmotic Dilators
Brief Title: Cervical Preparation for Same-Day Dilation & Evacuation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-45533
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Abortion, Second Trimester; Procedural Pain; Procedural Complication
Keywords: Cervical Dilation and Evacuation (D&E); Transcervical single-balloon catheter; Osmotic dilators; Adequate dilation; Patient satisfaction
MeSH Terms: conditions — Pain, Procedural; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a noninferiority parallel randomized control trial of two cervical preparation methods prior to same-day D&E.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcervical single-balloon catheter group (Experimental): Participants randomized to this arm will have cervical dilation done using a transcervical single-balloon catheter.
  Interventions: Device: Transcervical single-balloon catheter
- Osmotic dilators group (Active Comparator): Participants randomized to this arm will have cervical dilation done using osmotic dilators.
  Interventions: Device: Synthetic osmotic dilators

INTERVENTIONS:
Device: Transcervical single-balloon catheter — A single-balloon (Foley) catheter will be placed through the cervix and filled to 30cc of water or saline. The balloon will remain in the participant until their procedure, usually 3-4 hours, or earlier if it falls out on its own.
  Other Names: Foley catheter
  Arms: Transcervical single-balloon catheter group
Device: Synthetic osmotic dilators — Dilators will be maintained in the cervix between 3-4 hours, during which each dilator rod will swell several times its initial dried diameter.
  Other Names: Dilapan-S, seaweed laminaria
  Arms: Osmotic dilators group

SUMMARY:
This is a noninferiority randomized control trial of two cervical preparation methods prior to same-day Dilation & Evacuation (D&E). Cervical preparation is a process that softens and dilates the cervix prior to a procedure.

The primary objective is to evidence noninferiority of cervical preparation using a single-balloon catheter method when compared to a group receiving osmotic dilators, specifically in D&E operative time.

Secondary objectives will compare the two methods for adequate dilation, ability to complete the operation in the same day, participant pain, satisfaction and safety.

ELIGIBILITY:
Inclusion Criteria:

* Between 16 weeks 0 days - 18 weeks 6 days gestational age who are pursuing termination, based on reliable gestational age (defined as ultrasonography performed by a clinical provider, or a certain last menstrual period)
* Able to provide informed consent
* English- or Spanish-speaking
* Singleton intrauterine pregnancy

Exclusion Criteria:

* Allergy to betadine, aquacryl hydrogel, latex-free silicone single-balloon catheter, synthetic or natural osmotic dilators
* Fetal demise or known fetal anomaly
* BMI >45
* Incarceration or other inability to give informed consent
* Decide to undergo cervical preparation overnight prior to next-day D&E

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Dilation & Evacuation (D&E) Operative time | at end of procedure about 20 minutes
  the total duration in D&E operative time measured in minutes. Operative start time will be marked as the time that the speculum is inserted for the first time. Operative end time will be marked as the time that the speculum is removed at the end of the case.

SECONDARY OUTCOMES:
Participant preoperative pain | every hour until procedure, on average 3 hours
  Participant pain will be assessed via a 100 point visual analog scale immediately post-cervical preparation and at every hour interval until their D&E. Higher scores are associated with more pain.
Participant satisfaction | after dilation, on average 3 hours
  Participant satisfaction will be assessed with a 5-point Likert scale from very dissatisfied to very satisfied.
Cervical dilation | beginning of procedure, on average 3 hours
  Cervical dilation will be measured in millimeters at the beginning of the procedure by the surgeon.
Number of participants with adequate cervical dilation | beginning of procedure, on average 3 hours
  Abstracted from the operative record, dilation will be considered adequate if no manual dilation is needed.
Number of participants with surgery completed in the same day | 12 months
  Abstracted from the electronic medical record, whether the surgery was completed in the same day as the dilation will be recorded as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Anjanique Mariquit Lu, MD, Principal Investigator — Boston Medical Center, Obstetrics and Gynecology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No